CLINICAL TRIAL: NCT06986915
Title: Effect of Aerobic Exercise on Anthropometric, Biochemical, and Psychological Outcomes in Obese Adult Women: A Study at Dilla University, Ethiopia
Brief Title: Aerobic Exercise Effects on Health Indicators in Obese Women at Dilla University
Acronym: AEEHIOWDU
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Addisalem Girma (Other)
Collaborators: Dilla University (Other)
Responsible Party: Sponsor-Investigator, Addisalem Girma, A PhD Candidate, Mekelle University
Organization: Mekelle University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MUCNCS/PR134128/10ERC1383/2019
Record Dates: First submitted 2025-04-28; First posted 2025-05-23 (Actual); Last update posted 2025-05-23 (Actual); Status verified 2025-05

CONDITIONS: Obesity
Keywords: Obesity; Lipid profile; Body mass index; Aerobic exercise
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Intervention Model Description: Interventional Study Model: There is a single interventional cohort in which the participants engaged in an aerobic exercise program at a moderate intensity level alone without a control group.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Exercise group (Other): A participant group/Arm
  The arm of an obese adult woman is grouped as the Exercise group for the application of aerobic exercise intervention /treatment at a moderate intensity level.
  Interventions: Other: Aerobic exercise at moderate intensity level

INTERVENTIONS:
Other: Aerobic exercise at moderate intensity level — The intervention involved supervised aerobic activity sessions. Every session contained:
  Warm-up (5-10 minutes): To get the body ready, do some light stretching and low-intensity exercises.
  The primary aerobic activity (30-45 minutes) should consist of moderately intense exercises that aim to reach 60-75% of the participant's maximal heart rate.
  Cool-down (5-10 minutes): Stretching and a gradual decrease in activity to aid in recuperation.
  This intervention's objective was to evaluate how moderately intense aerobic exercise affected the anthropometric (body weight, BMI), biochemical (blood sugar, cholesterol), and psychological well-being indicators in obese adult women.

SUMMARY:
This clinical study examines how regular aerobic exercise affects the physical and mental health of obese adult women in Dilla, Ethiopia. Obesity is known to increase the risk of many health problems, including heart disease, diabetes, and emotional distress. Despite this, access to effective and affordable treatments can be limited in many low-resource settings. Physical activity, especially aerobic exercise like walking or jogging, is a simple and low-cost way to improve health. Still, more research is needed to understand its full benefits in specific populations.

The main goal of this study is to find out whether a structured aerobic exercise program can lead to improvements in three key areas:

Anthropometric measures, like weight, body mass index (BMI), and waist circumference.

Biochemical markers - including blood sugar (glucose), cholesterol levels, and other signs of metabolic health.

Psychological well-being - including symptoms of stress, depression, and overall mood.

The study involved obese adult women who met the inclusion criteria. Participants will be asked to engage in a supervised aerobic exercise program for twelve weeks. Measurements will be taken before and after the program to assess effects on the participants' physical and mental health.

This study postulates that regular aerobic exercise increased performance significantly in body composition, blood test results, and psychological health among obese women.

This research is expected to provide valuable evidence that shows exercise as a non-drug, low-cost intervention to help manage obesity and its related complications. This is especially important for communities like Dilla, where access to medical treatment may be limited, but lifestyle-based solutions can be both practical and effective.

DETAILED DESCRIPTION:
Obesity is characterized by an excessive accumulation of fat that interferes with the continual functioning of the body. Adequate body fat is necessary for maintaining health and proper bodily functions. Nevertheless, when fat surpasses normal levels and distributes throughout the body, it results in excessive fatness and obesity. These circumstances can hasten the onset of degenerative illnesses, present health challenges, and potentially reduce lifespans. The aim is to assess how twelve weeks of aerobic exercise impacts the anthropometric, biochemical, and psychological aspects among obese adult women. This research employed a quantitative methodology that involved a thorough and immersive research approach. Hence, a sampling frame was formed by a total of 70 obese adult women who were registered from the three campuses (main, Dilla referral hospital, and Odayaa'a) of Dilla University. The registered data/list was utilized to select participants through purposive sampling methods, and the researchers used this target population size as a Sampling frame. The BMI was the first general requirement used to classify the subjects as obese adult women. Next, 40 samples of obese adult women who met all major and relevant inclusion criteria were chosen from the sampling frame, which was created using the whole registered data/list of obese adult women. The sample size was determined by using the registered total female population information.

The BMI formula uses weight (in Kg or pounds) and height (in meters or inches) to form a simple calculation that results in a measure of your body fat. The formula for BMI was devised in the 1830s by Belgian mathematician Adolphe Quetelet and was universally expressed in kg/m2 (Alastair Hazell, 2020). It was calculated with the formulae,

BMI (Metric) = Weight in Kg / (Height in meters)2

This study aimed to evaluate the effect of aerobic exercise training on anthropometric, biochemical, and psychological outcomes in adult obese women. To achieve the this, 40 adult obese women (aged 30-38 years) were selected using a purposive sampling technique from Dilla University, Dilla, Ethiopia, who do not exercise regularly and were willing to participate in the exercise regime participate in this study. All participants were asked to abstain from taking pain-relieving medications (if any) until the exercise lasted (it was informed & consent was obtained from all participants before the baseline data was collected. Obese women who were contraindicated from doing exercise, physically disabled, breast feeders, and sick at the time of data collection were excluded as a general scanning from the study.

The anthropometric and psychological data were collected by the Principal Investigator, and the assistance with the follow-up of advisors. The Psychological questionnaires were adapted directly as it was prepared in English, then finalized and administered in the Amharic language, which is widely spoken in the city. Questions about socio-demographic characteristics were directly adopted from the standard Demographic and Health Survey (DHS) questionnaire (Central Statistical Agency of Ethiopia, 2011).

The procedure for blood biochemical parameters data, which is the experimental result for lipid profile (Total cholesterol (TC), High Density Lipoprotein (HDL), Low Density Lipoprotein (LDL), and Triglyceride) and fasting blood glucose test were measured in a calibrated biochemical analyzer at International clinical laboratory at Hawasa center.

Anthropometric measurements (Weight, BMI, triceps, suprailiac, & thigh skin folds, and waist circumference) were taken by using standardized equipment and standardized techniques. To minimize possible errors, measurements were made in duplicate by the same observer. Weight was measured using electronic weighing scales to the nearest 100 g. The scale was calibrated regularly, and the indicator was checked against zero reading before every measurement. Height was measured to the nearest 0.1 cm using a standing height board. Eventually, BMI (weight/height^2) was calculated, and obesity (BMI of 30-34.9 (Type I) & 35-40 (Type II)) was classified based on standard thresholds.

The present study was an experimental design with an interventional single-cohort design at the institutional level in obese adult women. For the study, 40 adult obese women were selected purposively from Dilla University, Dilla town, Ethiopia. Their ages range between 30 and 38 years. All selected subjects participated in the research voluntarily and cheerfully without any compulsion. The experimental group underwent the training for 12 weeks for 3 sessions per week (30 - 45 minutes), at a moderate intensity level, which was leveled/adjusted based on participants' (maximum heart rate). Pre-test & post-test were done for the blood biochemical parameters, but the anthropometric, psychological, and physiological variables were conducted four times at the end of each training month.

The study implemented a 30 - 45 minute aerobic exercise intervention, which included various exercises such as on spot marching, marching with side up and down arm movement, side to side movement, side to side with bending knees, side step and kick, double side step and kick, forward marching with arm swing, V step movement, and zig-zag forward movement. Before the exercise session, there was a 5-minute period to ensure the readiness and safety of the participants, followed by a 5-minute warm-up exercise. Additionally, a 5-minute cool-down exercise was performed after the aerobic exercises. Following the exercise session, there was a 10-minute period dedicated to discussion and feedback. Finally, there was a 5-minute allowance for any time wasted during the session to be compensated; the exercise regimen consisted of a frequency of three times per week on nonconsecutive days. The intensity level was set at 50-60% of maximum effort, which is considered moderate for the targeted age group. The exercise protocol involved four sets with six repetitions each. Rest periods of 30 seconds were provided between exercises, while 10 seconds were allowed between sets. The researchers, with Dilla University Community Gym (DUCG) professionals, define these guidelines.

Intensity of the exercise was determined by the subjects' maximum heart rates, which were measured using the L8-R8 Smart Heart Rate Wristband, Shenzhen L8star Technology Co., Ltd, China. This confirmed that a standard intensity level suitable for healthy individuals with a heart rate ranging from 57 to 75 beats per minute was selected to set the training intensity. The aim was to maintain a consistent exercise intensity level with the biological characteristics of the age group, as defined by the World Health Organization (WHO).

The analysis was performed using the SPSS program (IBM SPSS Statistics version 20, IBM, USA). Demographic information of the participants was displayed using frequencies and percentages. When dealing with continuous variables that displayed a normal distribution, group differences were assessed using t-tests and one-way ANOVA. In cases where the distribution deviated from normality, the Mann-Whitney test was utilized. The normality of the data was evaluated in histograms, standard Q-Q plots, and the Kolmogorov-Smirnov test. To explore multiple comparisons between paired treatments, the Bonferroni tests (which included the LSD test, Duncan's test, and Tukey's test) were employed.

This research investigated how aerobic exercise influences various aspects of health in obese adult women enrolled at Dilla University in Ethiopia. The primary aim was to examine whether engaging in moderate-intense aerobic activity could improve physical, biochemical, and psychological health outcomes.

To achieve this, the study focused on three key areas:

Anthropometric (Physical) Changes: Researchers recorded body measurements such as weight, body mass index (BMI), waist circumference, and other indicators of body composition. These measurements helped determine the physical effects of exercise, such as weight loss or changes in body shape.

Biochemical Variables: Blood samples were analyzed to monitor important biochemical markers, including cholesterol levels, blood glucose, and other metabolic indicators. These values provided insight into how aerobic exercise might reduce health risks related to obesity, such as heart disease and diabetes.

Psychological Well-being: The study also evaluated mental health factors such as anxiety, self-esteem, and body satisfaction. By using standardized psychological assessments, researchers assessed whether participation in aerobic exercise contributed to improved mental well-being and reduced symptoms of psychological distress.

Participants underwent a structured aerobic exercise program for 12 weeks, and their health status was measured both before and after the intervention. By comparing the results, the study aimed to determine the effectiveness of aerobic exercise in promoting overall health among obese women.

In summary, the study provided evidence on how regular aerobic activity can positively affect the body, internal health markers, and psychological state, supporting its role as a valuable intervention for managing obesity and enhancing quality of life.

ELIGIBILITY:
Inclusion Criteria:

* women working at Dilla University
* age ranged from 30 to 38 years
* obese women (BMI ≥ 30 kg/m2)
* did not engage in regular exercise
* willing to participate in the study

Exclusion Criteria:

* women with chronic disease
* lifetime tablet
* Not willing to the blood sampling
* Irregular presence for the intervention
* Sergery less than a year

Ages: 30 Years to 38 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2019-12-05 (Actual); Primary Completion 2020-02-11 (Actual); Study Completion 2020-05-16 (Actual)

PRIMARY OUTCOMES:
Anthropometric Outcome Measures | 6 Months
  Outcome measure:
  Triceps thickness in millimeters.
  Measure description -
  The skinfold thickness at this site was measured three times using a caliper, and the average of the three readings was recorded. This site is one of several used to estimate overall body fat percentage.
  Outcome measure -
  Suprailiac thickness in millimeters.
  Measure description -
  The skinfold thickness at this site was measured three times using a caliper, and the average of the three readings was recorded. This site is one of several used to estimate overall body fat percentage.
  Outcome measure -
  Thigh thickness in millimeters.
  Measure descriptions -
  The skinfold thickness at this site was measured three times using a caliper, and the average of the three readings was recorded. This site is one of several used to estimate overall body fat percentage.
  Additional explanation is found in the detailed Description.

SECONDARY OUTCOMES:
Biochemical Outcome Measures | 6 Months
  Outcome Measure - Total cholesterol (TC) in milligrams per deciliter. Measure description - A 5 ml blood sample is taken and then tested by an automatic blood analyzer. Outcome measure - High Density Lipoprotein (HDL)in milligrams per deciliter. Measure description - A 5 ml blood sample is taken, then tested by an automatic blood analyzer. Outcome Measure - Low Density Lipoprotein (LDL) in milligrams per deciliter. Measure description - A 5 ml blood sample is taken, then tested by an automatic blood analyzer. Triglyceride in miligrams per deciliter. Measure description - A 5 ml blood sample is taken and then tested by an automatic blood analyzer. Outcome measure - Fasting blood Glucose (FBG) in milligrams per deciliter. Measure description - A small handheld device, known as a glucose meter or glucometer, is used to measure sugar (glucose) in a blood sample. Typically, a drop of blood obtained through a finger prick on an empty stomach is sufficient for analysis using a test strip.

CONTACTS AND LOCATIONS:
Locations (1):
- Dilla University, Awasa, Southern Ethiopia, Ethiopia

IPD SHARING:
Plan to Share IPD: No
The sponsor owns the data and uses it exclusively for internal research.

REFERENCES:
- [Background] Stepien A, Stepien M, Wlazel RN, Paradowski M, Banach M, Rysz J. Assessment of the relationship between lipid parameters and obesity indices in non-diabetic obese patients: a preliminary report. Med Sci Monit. 2014 Dec 16;20:2683-8. doi: 10.12659/MSM.890845. PMID 25512170
- [Background] Lee S, Kuk JL, Davidson LE, Hudson R, Kilpatrick K, Graham TE, Ross R. Exercise without weight loss is an effective strategy for obesity reduction in obese individuals with and without Type 2 diabetes. J Appl Physiol (1985). 2005 Sep;99(3):1220-5. doi: 10.1152/japplphysiol.00053.2005. Epub 2005 Apr 28. PMID 15860689
- [Background] Slentz CA, Houmard JA, Johnson JL, Bateman LA, Tanner CJ, McCartney JS, Duscha BD, Kraus WE. Inactivity, exercise training and detraining, and plasma lipoproteins. STRRIDE: a randomized, controlled study of exercise intensity and amount. J Appl Physiol (1985). 2007 Aug;103(2):432-42. doi: 10.1152/japplphysiol.01314.2006. Epub 2007 Mar 29. PMID 17395756
- [Background] Ballor DL, Katch VL, Becque MD, Marks CR. Resistance weight training during caloric restriction enhances lean body weight maintenance. Am J Clin Nutr. 1988 Jan;47(1):19-25. doi: 10.1093/ajcn/47.1.19. PMID 3337037
- [Background] 5. Nikseresht, A., & Sarreshtedari, S. (2016). The effect of 8-week aerobic exercise on body composition and lipid profile in overweight women. International Journal of Medical Research & Health Sciences, 5(4), 121-126.
- [Background] 4. Alizadeh, L., Moghaddam Tabrizi, F., & Salehi, F. (2014). Effects of aerobic exercise on body composition and lipid profile in overweight women. Journal of Family & Reproductive Health, 8(2), 77-82.
- [Background] Dieli-Conwright CM, Courneya KS, Demark-Wahnefried W, Sami N, Lee K, Sweeney FC, Stewart C, Buchanan TA, Spicer D, Tripathy D, Bernstein L, Mortimer JE. Aerobic and resistance exercise improves physical fitness, bone health, and quality of life in overweight and obese breast cancer survivors: a randomized controlled trial. Breast Cancer Res. 2018 Oct 19;20(1):124. doi: 10.1186/s13058-018-1051-6. PMID 30340503
- [Background] de Freitas RW, de Araujo MF, Lima AC, Pereira DC, Alencar AM, Damasceno MM. Study of lipid profile in a population of university students. Rev Lat Am Enfermagem. 2013 Sep-Oct;21(5):1151-8. doi: 10.1590/S0104-11692013000500019. English, Portuguese, Spanish. PMID 24142225
- [Background] Vatansev, H. (2014). The effects of 8-week aerobic exercises on the blood lipid and body composition of the owerweight and obese females the effects of 8-week aerobic exercises on the blood lipid and body composition of the owerweight and obese females. January 2010.
- [Background] Stephens JM. The fat controller: adipocyte development. PLoS Biol. 2012;10(11):e1001436. doi: 10.1371/journal.pbio.1001436. Epub 2012 Nov 27. PMID 23209380
- [Background] Nuttall FQ. Body Mass Index: Obesity, BMI, and Health: A Critical Review. Nutr Today. 2015 May;50(3):117-128. doi: 10.1097/NT.0000000000000092. Epub 2015 Apr 7. PMID 27340299
- [Background] Alizadeh Z, Halabchi F, Bodaghabadi Z, Zarandi MM, Abolhasani M, Seifi V, Khazaei R, Ghanadi S, Mazaheri R, Tabesh MR. Non-invasive Body Contouring Technologies: An Updated Narrative Review. Aesthetic Plast Surg. 2024 Feb;48(4):659-679. doi: 10.1007/s00266-023-03647-x. Epub 2023 Sep 25. PMID 37749418
- [Background] Ross R, Dagnone D, Jones PJ, Smith H, Paddags A, Hudson R, Janssen I. Reduction in obesity and related comorbid conditions after diet-induced weight loss or exercise-induced weight loss in men. A randomized, controlled trial. Ann Intern Med. 2000 Jul 18;133(2):92-103. doi: 10.7326/0003-4819-133-2-200007180-00008. PMID 10896648
- See also: Related articles — https://www.ncbi.nlm.nih.gov/pmc/articles/PMC4744305/